CLINICAL TRIAL: NCT04102189
Title: Effect and Safety of Semaglutide 2.4 mg Once Weekly on Weight Management in Adolescents With Overweight or Obesity
Brief Title: A Research Study on How Well Semaglutide Works in Adolescents With Overweight or Obesity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9536-4451; U1111-1215-7560 (Other: World Health Organization (WHO)); 2018-002431-18 (EudraCT Number)
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Results first posted 2023-04-18 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Semaglutide (Experimental): 2.4 mg or maximum tolerated dose (MTD) injected subcutaneously (under the skin, s.c.) once weekly
  Interventions: Drug: Semaglutide
- Placebo (Placebo Comparator): Placebo injected s.c. once weekly .
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Semaglutide — Participants will receive semaglutide s.c. once weekly for a dose escalation period of 16 weeks and a maintenance period of 52 weeks
  Arms: Semaglutide
Other: Placebo — Participants will receive semaglutide placebo s.c. once weekly for a total of 68 weeks
  Arms: Placebo

SUMMARY:
This study will look at the change in teenagers' body weight from the start to the end of the study. This is to compare the effect on body weight in teenagers taking semaglutide (a new medicine) and teenagers taking "dummy" medicine. The teenagers in the study and their parents will also have talks with study staff about healthy food choices, how to be more physically active and what they can do to help the teenagers lose weight. The teenagers will either get semaglutide or "dummy" medicine - which treatment is decided by chance. The teenagers will take 1 injection every week, on the same day of the week for about 15 months. The study medicine is injected with a thin needle in a skin fold in the stomach, thigh or upper arm. The teenagers will have 17 clinic visits, will have blood samples taken and will have to complete questionnaires and keep a diary. All this will be explained before study start.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent of parent(s) or legally acceptable representative of subject and child assent, as appropriate obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
* Male or female, ages 12 to below 18 years at the time of signing informed consent
* BMI equal to or above 95th percentile OR equal to or above 85th percentile (on gender and age-specific growth charts (CDC.gov)) with 1 or more weight related comorbidity (treated or untreated): hypertension, dyslipidaemia, obstructive sleep apnoea or type 2 diabetes
* History of at least one self-reported unsuccessful dietary effort to lose weight

For subjects with type 2 diabetes at screening the following inclusion criteria apply in addition:

- HbA1c equal to or below 10.0% (86 mmol/mol) as measured by central laboratory at screening

Exclusion Criteria:

* Prepubertal subjects (Tanner stage 1)
* History of type 1 diabetes
* A self-reported (or by parent(s)/legally acceptable representative where applicable) change in body weight above 5 kg (11 lbs) within 90 days before screening irrespective of medical records
* Subjects with secondary causes of obesity (i.e., hypothalamic, monogenic or endocrine causes)
* For subjects with type 2 diabetes only: Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within the past 90 days prior to screening. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 201 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (51):
- United States (23):
  - Children's Hospital Los Angeles - Endocrinology, Los Angeles, California
  - Solaris Clinical Research, Meridian, Idaho
  - Pennington Biomed Res Ctr, Baton Rouge, Louisiana
  - DelRicht Research, Gretna, Louisiana
  - Barry J. Reiner, MD LLC, Baltimore, Maryland
  - Massachusetts General Hospital_Cary, Boston, Massachusetts
  - University of Minnesota_CPOM, Minneapolis, Minnesota
  - University of Minnesota_Minneapolis, Minneapolis, Minnesota
  - UBMD Peds-Div of Endo/Diabetes, Buffalo, New York
  - WakeMed Childn Endo-Dbt_Raleig, Raleigh, North Carolina
  - Valley Weight Loss Clinic, Fargo, North Dakota
  - Aventiv Research Inc, Columbus, Ohio
  - PriMed Clinical Research, Dayton, Ohio
  - Geisinger Clinic, Danville, Pennsylvania
  - Children's Hosptl Philadelphia, Philadelphia, Pennsylvania
  - UPMC Child Hosp-Pittsburgh, Pittsburgh, Pennsylvania
  - Medical Research South, LLC_Cary, Goose Creek, South Carolina
  - Greenville Hospital System Pediatric Endo, Greenville, South Carolina
  - Monument Health Clinical Rsrch, Rapid City, South Dakota
  - Discovery MM Services, Inc, Houston, Texas
  - Univ Of Texas Hlth Science Cntr, San Antonio, Texas
  - National Clin Res Inc., Richmond, Virginia
  - Marshfield Clinic, Marshfield, Wisconsin
- Austria (3):
  - Fließer-Görzer [Ordination], Saint Stefan
  - Universitätsklinik für Kinder und Jugendheilkunde Haus E, Salzburg
  - Ordination Dr. Hanusch, Vienna
- Belgium (4):
  - UZ Brussel, Brussels
  - Cliniques Universitaires Saint-Luc - Serv. Pédiatrie, Brussels
  - UZA - UZ Antwerpen - Kinderziekenhuis, Edegem
  - UZ Leuven - Kindergeneeskunde, Leuven
- Croatia (3):
  - Klinički bolnički centar Rijeka, pedijatrija, Rijeka
  - KBC "Sestre Milosrdnice", Zagreb
  - KBC Zagreb, Zavod za dječju endokrinologiju i dijabetes, Zagreb
- Ireland (4):
  - Clinical Research Centre, St. Vincent's University Hospital,, Dublin, Leinster
  - CHI Crumlin Dept of Endocrinology, Dublin
  - CRF HRB - Galway, Galway
  - Wexford General Hospital - UCD CRC, Wexford
- Consultorio de Endocrinología y Pediatría, Puebla City, Mexico
- Russia (7):
  - Republic Children's Hospital of Ministry of Health of Udmurt, Izhevsk
  - RMAPE, Moscow
  - NSMU paediatric clinic, Novosibirsk
  - FSBEI of Higher Education "Rostov State Medical University", Rostov-on-Don
  - City Children Endocrinology Center n.a. Raukhfus, Saint Petersburg
  - SPSBHI City Children out-patient clinic #44, Saint Petersburg
  - Siberian State Medical University, Tomsk
- United Kingdom (6):
  - Clifton Medical Centre, Rotherham, South Yorkshire
  - Birmingham Children's Hospital, Birmingham
  - University Hospitals Bristol & Weston NHS Foundation Trust, Bristol
  - University College Hospital Hospital - Paediatric Services, London
  - Ecclesfield Group Practice, Sheffield
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Result] Weghuber D, Barrett T, Barrientos-Perez M, Gies I, Hesse D, Jeppesen OK, Kelly AS, Mastrandrea LD, Sorrig R, Arslanian S; STEP TEENS Investigators. Once-Weekly Semaglutide in Adolescents with Obesity. N Engl J Med. 2022 Dec 15;387(24):2245-2257. doi: 10.1056/NEJMoa2208601. Epub 2022 Nov 2. PMID 36322838
- [Derived] Kelly AS, Arslanian S, Hesse D, Iversen AT, Korner A, Schmidt S, Sorrig R, Weghuber D, Jastreboff AM. Reducing BMI below the obesity threshold in adolescents treated with once-weekly subcutaneous semaglutide 2.4 mg. Obesity (Silver Spring). 2023 Aug;31(8):2139-2149. doi: 10.1002/oby.23808. Epub 2023 Jul 9. PMID 37196421
- [Derived] Weghuber D, Boberg K, Hesse D, Jeppesen OK, Sorrig R, Kelly AS; STEP TEENS Investigators. Semaglutide treatment for obesity in teenagers: a plain language summary of the STEP TEENS research study. J Comp Eff Res. 2023 Feb;12(2):e220187. doi: 10.2217/cer-2022-0187. Epub 2022 Dec 19. PMID 36534451
- [Derived] Cuda S, Censani M. Progress in pediatric obesity: new and advanced therapies. Curr Opin Pediatr. 2022 Aug 1;34(4):407-413. doi: 10.1097/MOP.0000000000001150. Epub 2022 Jul 5. PMID 35797460

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 37 sites in 8 countries, as follows: Austria (3), Belgium (4), Croatia (3), Ireland (1), Mexico (1), Russia (7), Great Britain (6), United States (12).
Pre-assignment Details: Participants were randomized 2:1 to receive either semaglutide subcutaneously (s.c.) once weekly or semaglutide placebo s.c. once weekly for a dose escalation period of 16 weeks and a maintenance period of 52 weeks. This was followed by a 7-week follow-up period after 'end of treatment' due to the long half-life of semaglutide.
Groups:
- Semaglutide 2.4 mg: Participants received once weekly s.c. injection of semaglutide for 68 weeks. Participants initially received 0.25 milligrams (mg) of semaglutide and the dose was then escalated once in 4 weeks for 16 weeks until the target dose of 2.4 mg was reached which was maintained for a period of 52 weeks: 0.25 mg (week 1 to week 4), 0.5 mg (week 5 to week 8), 1.0 mg (week 9 to week 12), 1.7 mg (week 13 to week 16) and 2.4 mg (week 17 to week 68). The treatment was an adjunct to a reduced-calorie diet and increased physical activity.
- Placebo: Participants received once weekly s.c. injection of placebo matched to semaglutide for 68 weeks. The treatment was an adjunct to a reduced-calorie diet and increased physical activity.
Period: Overall Study
Arm/Group | Semaglutide 2.4 mg | Placebo
Started | 134 | 67
Treated | 133 | 67
Full Analysis Set (FAS) | 134 | 67
Safety Analysis Set | 133 | 67
Completed | 132 | 64
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Withdrawal by parent/guardian | 0 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomized participants according to the intention-to-treat principle.
Groups:
- Total: Total of all reporting groups
Arm/Group | Semaglutide 2.4 mg | Placebo | Total
Number analyzed (Participants) | 134 | 67 | 201
Age, Continuous [Mean (Standard Deviation); unit: Years] | 15.5 (1.5) | 15.3 (1.6) | 15.4 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 41 | 125
  Male | 50 | 26 | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 8 | 22
  Not Hispanic or Latino | 120 | 59 | 179
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 104 | 55 | 159
  Race: Other | 14 | 6 | 20
  Race: Black or African American | 11 | 5 | 16
  Race: Asian | 3 | 1 | 4
  Race: American Indian or Alaska Native | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Mass Index (BMI) (Percentage [%])
Description: Change in BMI (%) from baseline to week 68 is presented. Data is reported for 'in-trial' period: the uninterrupted time interval from randomization to last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: The full analysis set (FAS) included all randomized participants according to the intention-to-treat principle. Overall Number of Participants Analyzed = number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage change of BMI
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 131 | 62
Percentage change of BMI | -16.2 (12.9) | -0.1 (8.6)
Statistical Analysis 1: Comparison: Semaglutide 2.4 mg vs Placebo; Responses were analyzed using an analysis of covariance model with randomized treatment, stratification groups (sex and Tanner stage at baseline) and the interaction between stratification groups as factors and baseline BMI as covariate; Test type: Superiority; p < .0001, ANCOVA; Treatment difference = -16.75, 95% CI 2-sided [-20.27 to -13.23]

2. Secondary Outcome: Percentage of Participants Achieving Greater Than or Equal to (>=) 5% Reduction of Body Weight (Yes/no)
Description: Percentage of participants who achieved >= 5% weight reduction from baseline (week 0) to week 68 is presented. In the reported data, 'Yes' infers the percentage of participants who have achieved >= 5% weight reduction, whereas 'No' infers the percentage of participants who did not achieve >= 5% weight reduction. Data is reported for 'in-trial' period: the uninterrupted time interval from date of randomization to last contact with trial site.
Time Frame: At week 68
Population: FAS included all randomized participants according to the intention-to-treat principle. Overall Number of Participants Analyzed = number of participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 131 | 62
Percentage of participants
  Yes | 72.5 | 17.7
  No | 27.5 | 82.3

3. Secondary Outcome: Change in Body Weight (Kilograms [kg])
Description: Change in body weight (kg) from baseline to week 68 is presented. Data is reported for 'in-trial' period: the uninterrupted time interval from randomization to last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 131 | 62
kg | -15.7 (14.6) | 2.3 (9.7)

4. Secondary Outcome: Change in Body Weight (%)
Description: Change in body weight (%) from baseline to week 68 is presented. Data is reported for 'in-trial' period: the uninterrupted time interval from randomization to last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage change of body weight
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 131 | 62
Percentage change of body weight | -14.8 (13.2) | 2.3 (9.1)

5. Secondary Outcome: Percentage of Participants Achieving >=10% Reduction of Body Weight (Yes/no)
Description: Percentage of participants who achieved >= 10% weight reduction from baseline (week 0) to week 68 is presented. In the reported data, 'Yes' infers the percentage of participants who have achieved >= 10% weight reduction, whereas 'No' infers the percentage of participants who did not achieve >= 10% weight reduction. Data is reported for 'in-trial' period: the uninterrupted time interval from date of randomization to last contact with trial site.
Time Frame: At week 68
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 131 | 62
Percentage of participants
  Yes | 61.8 | 8.1
  No | 38.2 | 91.9

6. Secondary Outcome: Percentage of Participants Achieving >=15% Reduction of Body Weight (Yes/no)
Description: Percentage of participants who achieved >= 15% weight reduction from baseline (week 0) to week 68 is presented. In the reported data, 'Yes' infers the percentage of participants who have achieved >= 15% weight reduction, whereas 'No' infers the percentage of participants who did not achieve >= 15% weight reduction. Data is reported for 'in-trial' period: the uninterrupted time interval from date of randomization to last contact with trial site.
Time Frame: At week 68
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 131 | 62
Percentage of participants
  Yes | 53.4 | 4.8
  No | 46.6 | 95.2

7. Secondary Outcome: Percentage of Participants Achieving >=20% Reduction of Body Weight (Yes/no)
Description: Percentage of participants who achieved >= 20% weight reduction from baseline (week 0) to week 68 is presented. In the reported data, 'Yes' infers the percentage of participants who have achieved >= 20% weight reduction, whereas 'No' infers the percentage of participants who did not achieve >= 20% weight reduction. Data is reported for 'in-trial' period: the uninterrupted time interval from date of randomization to last contact with trial site.
Time Frame: At week 68
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 131 | 62
Percentage of participants
  Yes | 37.4 | 3.2
  No | 62.6 | 96.8

8. Secondary Outcome: Change in BMI Percentage of the 95th Percentile on Gender and Age-specific Growth Charts (CDC.Gov [CDC: {Centers for Disease Control and Prevention}])
Description: Change from baseline in BMI percentage of the 95th percentile on gender and age-specific growth charts (CDC.gov) at week 68 is presented. CDC gender and age-specific growth charts: normal (BMI less than [<] 85th percentile), overweight (BMI greater than or equal to [>=] 85th - <95th percentile), obesity class I (BMI >=95th - <120% of the 95th percentile), obesity class II (BMI >=120% of the 95th percentile - <140% of the 95th percentile) and obesity class III (BMI >=140% of the 95th percentile). Data is reported for 'in-trial' period: the uninterrupted time interval from randomization to last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage point of BMI
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 131 | 62
Percentage point of BMI | -24.9 (17.0) | -4.5 (10.5)

9. Secondary Outcome: Percentage of Participants Achieving Improvement in Weight Category (Yes/no)
Description: Percentage of participants who achieved improvement in weight category from baseline (week 0) to week 68 is presented. Improvement in weight category was defined as being in a lower weight category at week 68 compared to baseline according to CDC gender and age-specific growth charts: normal (BMI <85th percentile), overweight (BMI >=85th - <95th percentile), obesity class I (BMI >=95th - <120% of the 95th percentile), obesity class II (BMI >=120% of the 95th percentile - <140% of the 95th percentile) and obesity class III (BMI >=140% of the 95th percentile). In the reported data, 'Yes' infers the percentage of participants who have achieved improvement in weight category, whereas 'No' infers the percentage of participants who did not achieve improvement in weight category. Data is reported for 'in-trial' period: the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: At week 68
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 131 | 62
Percentage of participants
  Yes | 71.8 | 21.0
  No | 28.2 | 79.0

10. Secondary Outcome: Change in BMI (Standard Deviation Score [SDS])
Description: Change in BMI SDS from baseline to week 68 is presented. The SDS scores are also called as z-scores. BMI SDS was calculated using the following formula: Z=[(value /M)^L - 1] / S*L; where L, M and S are median (M), skewness (L) and variation coefficient (S) of children/adolescents' BMI provided for each sex and age. For each subject, a standard deviation score Z (SDS) was calculated based on age and sex referring to the values L, M and S. The method is described in the world health organisation (WHO) Multicentre Growth Reference, which also contains the values for L, M and S by age and sex. For Z (SDS) scores below -3 and above 3, the score was adjusted as described in the WHO instruction. Possible values range from -3 to +3, a negative score being beneficial. Data is reported for 'in-trial' period: the uninterrupted time interval from randomization to last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: standard deviation score
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 131 | 62
standard deviation score | -1.1 (0.9) | -0.1 (0.5)

11. Secondary Outcome: Change in BMI (Kilograms Per Meter Square [kg/m^2])
Description: Change in BMI (kg/m^2) from baseline to week 68 is presented. Data is reported for 'in-trial' period: the uninterrupted time interval from randomization to last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 131 | 62
kg/m^2 | -5.9 (4.9) | 0.0 (3.1)

12. Secondary Outcome: Change in Waist Circumference
Description: Change in waist circumference (centimeters [cm]) from baseline to week 68 is presented. Data is reported for 'in-trial' period: the uninterrupted time interval from randomization to last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 131 | 62
cm | -12.7 (12.2) | -0.5 (6.5)

13. Secondary Outcome: Percentage of Participants Achieving >=5% Reduction of BMI (Yes/no)
Description: Percentage of participants who achieved >= 5% reduction of BMI from baseline (week 0) to week 68 is presented. In the reported data, 'Yes' infers the percentage of participants who have achieved >= 5% BMI reduction, whereas 'No' infers the percentage of participants who did not achieve >= 5% BMI reduction. Data is reported for 'in-trial' period: the uninterrupted time interval from date of randomization to last contact with trial site.
Time Frame: At week 68
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 131 | 62
Percentage of participants
  Yes | 75.6 | 22.6
  No | 24.4 | 77.4

14. Secondary Outcome: Change in Systolic Blood Pressure
Description: Change in systolic blood pressure from baseline to week 68 is presented. Data is reported for 'in-trial' period: the uninterrupted time interval from randomization to last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 131 | 62
millimeters of mercury (mmHg) | -3 (12) | -1 (9)

15. Secondary Outcome: Change in Diastolic Blood Pressure
Description: Change in diastolic blood pressure from baseline to week 68 is presented. Data is reported for 'in-trial' period: the uninterrupted time interval from randomization to last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 131 | 62
mmHg | -2 (9) | -1 (8)

16. Secondary Outcome: Change in Glycated Haemoglobin (HbA1c) (%)
Description: Change in HbA1c (%) from baseline to week 68 is presented. Data is reported for 'in-trial' period: the uninterrupted time interval from randomization to last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 126 | 59
Percentage of HbA1c | -0.4 (0.3) | -0.1 (0.3)

17. Secondary Outcome: Change in HbA1c (Millimoles Per Mole [mmol/Mol])
Description: Change in HbA1c (mmol/mol) from baseline to week 68 is presented. Data is reported for 'in-trial' period: the uninterrupted time interval from randomization to last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 126 | 59
mmol/mol | -4.2 (3.5) | -1.2 (2.9)

18. Secondary Outcome: Change in Fasting Plasma Glucose (Millimoles Per Liter [mmol/L])
Description: Change in fasting plasma glucose (mmol/L) from baseline to week 68 is presented. Data is reported for 'in-trial' period: the uninterrupted time interval from randomization to last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 127 | 57
mmol/L | -0.2 (0.5) | 0.0 (0.5)

19. Secondary Outcome: Change in Fasting Plasma Glucose (Milligrams Per Deciliter [mg/dL])
Description: Change in fasting plasma glucose (mg/dL) from baseline to week 68 is presented. Data is reported for 'in-trial' period: the uninterrupted time interval from randomization to last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 127 | 57
mg/dL | -4.2 (9.6) | 0.0 (8.6)

20. Secondary Outcome: Change in Fasting Insulin (Picomoles Per Liter [Pmol/L]): Ratio to Baseline
Description: Change in fasting insulin (pmol/L) from baseline to week 68 is presented as ratio to baseline. Data is reported for 'in-trial' period: the uninterrupted time interval from randomization to last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting insulin
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 120 | 51
Ratio of fasting insulin | 0.64 (62.9) | 0.99 (58.2)

21. Secondary Outcome: Change in Fasting Insulin (Milli International Units Per Milliliter [mIU/mL]): Ratio to Baseline
Description: Change in fasting insulin (mIU/mL) from baseline to week 68 is presented as ratio to baseline. Data is reported for 'in-trial' period: the uninterrupted time interval from randomization to last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting insulin
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 120 | 51
Ratio of fasting insulin | 0.64 (62.9) | 0.99 (58.2)

22. Secondary Outcome: Change in Total Cholesterol (mmol/L): Ratio to Baseline
Description: Change in total cholesterol (mmol/L) from baseline to week 68 is presented as ratio to baseline. Data is reported for 'in-trial' period: the uninterrupted time interval from randomization to last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total cholesterol
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 130 | 58
Ratio of total cholesterol | 0.92 (14.6) | 0.98 (9.4)

23. Secondary Outcome: Change in Total Cholesterol (mg/dL): Ratio to Baseline
Description: Change in total cholesterol (mg/dL) from baseline to week 68 is presented as ratio to baseline. Data is reported for 'in-trial' period: the uninterrupted time interval from randomization to last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total cholesterol
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 130 | 58
Ratio of total cholesterol | 0.92 (14.6) | 0.98 (9.4)

24. Secondary Outcome: Change in High-density Lipoprotein (HDL) Cholesterol (mmol/L): Ratio to Baseline
Description: Change in HDL cholesterol (mmol/L) from baseline to week 68 is presented as ratio to baseline. Data is reported for 'in-trial' period: the uninterrupted time interval from randomization to last contact with trial site.
Time Frame: Baseline (week 0), week 68:
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HDL cholesterol
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 124 | 57
Ratio of HDL cholesterol | 1.08 (17.5) | 1.03 (21.5)

25. Secondary Outcome: Change in High-density Lipoprotein (HDL) Cholesterol (mg/dL): Ratio to Baseline
Description: Change in HDL cholesterol (mg/dL) from baseline to week 68 is presented as ratio to baseline. Data is reported for 'in-trial' period: the uninterrupted time interval from randomization to last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HDL cholesterol
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 124 | 57
Ratio of HDL cholesterol | 1.08 (17.5) | 1.03 (21.5)

26. Secondary Outcome: Change in Low-density Lipoprotein (LDL) Cholesterol (mmol/L): Ratio to Baseline
Description: Change in LDL cholesterol (mmol/L) from baseline to week 68 is presented as ratio to baseline. Data is reported for 'in-trial' period: the uninterrupted time interval from randomization to last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of LDL cholesterol
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 129 | 58
Ratio of LDL cholesterol | 0.91 (20.9) | 0.96 (15.4)

27. Secondary Outcome: Change in LDL Cholesterol (mg/dL): Ratio to Baseline
Description: Change in LDL cholesterol (mg/dL) from baseline to week 68 is presented as ratio to baseline. Data is reported for 'in-trial' period: the uninterrupted time interval from randomization to last contact with trial site.
Time Frame: Baseline (week 0), week 68:
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of LDL cholesterol
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 129 | 58
Ratio of LDL cholesterol | 0.91 (20.9) | 0.96 (15.4)

28. Secondary Outcome: Change in Very Low-density Lipoprotein (VLDL) Cholesterol (mmol/L): Ratio to Baseline
Description: Change in VLDL cholesterol (mmol/L) from baseline to week 68 is presented as ratio to baseline. Data is reported for 'in-trial' period: the uninterrupted time interval from randomization to last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of VLDL cholesterol
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 129 | 58
Ratio of VLDL cholesterol | 0.71 (46.1) | 1.03 (40.8)

29. Secondary Outcome: Change in VLDL Cholesterol (mg/dL): Ratio to Baseline
Description: Change in VLDL cholesterol (mg/dL) from baseline to week 68 is presented as ratio to baseline. Data is reported for 'in-trial' period: the uninterrupted time interval from randomization to last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of VLDL cholesterol
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 129 | 58
Ratio of VLDL cholesterol | 0.71 (46.1) | 1.03 (40.8)

30. Secondary Outcome: Change in Triglycerides (mmol/L): Ratio to Baseline
Description: Change in triglycerides (mmol/L) from baseline to week 68 is presented as ratio to baseline. Data is reported for 'in-trial' period: the uninterrupted time interval from randomization to last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of triglycerides
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 129 | 58
Ratio of triglycerides | 0.71 (45.8) | 1.04 (40.9)

31. Secondary Outcome: Change in Triglycerides (mg/dL): Ratio to Baseline
Description: Change in triglycerides (mg/dL) from baseline to week 68 is presented as ratio to baseline. Data is reported for 'in-trial' period: the uninterrupted time interval from randomization to last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of triglycerides
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 129 | 58
Ratio of triglycerides | 0.71 (45.8) | 1.04 (40.9)

32. Secondary Outcome: Change in Alanine Aminotransferase (ALT): Ratio to Baseline
Description: Change in ALT (units per liter [U/L]) from baseline to week 68 is presented as ratio to baseline. Data is reported for 'in-trial' period: the uninterrupted time interval from randomization to last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of ALT
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 128 | 58
Ratio of ALT | 0.79 (63.8) | 1.00 (44.3)

33. Secondary Outcome: Number of Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical trial participant administered or using a medicinal product, whether or not considered related to the medicinal product or usage. All AEs reported here are TEAEs. TEAE is defined as an event that had onset date during the on-treatment period. The on-treatment period was defined as the interval from first to last trial product administration plus 7 weeks of follow-up and excluding any period of temporary treatment interruption defined as greater than (>) 7 consecutive missed doses (corresponding to >7 weeks off-treatment).
Time Frame: From baseline (week 0) to week 75
Population: The safety analysis set (SAS) included all randomized participants exposed to at least one dose of randomized treatment.
Measure: Number; unit: Events
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 133 | 67
Events | 792 | 328

34. Secondary Outcome: Number of Treatment-emergent Serious Adverse Events (SAEs)
Description: An SAE is an AE that fulfils at least one of the following criteria: 1) results in death; 2) is life-threatening; 3) requires inpatient hospitalisation or prolongation of existing hospitalisation; 4) results in persistent disability/incapacity; 5) is a congenital anomaly/birth defect; 6) important medical event. All AEs reported here are TEAEs. TEAE is defined as an event that had onset date during the on-treatment period. The on-treatment period was defined as the interval from first to last trial product administration plus 7 weeks of follow-up and excluding any period of temporary treatment interruption defined as >7 consecutive missed doses (corresponding to >7 weeks off-treatment).
Time Frame: From baseline (week 0) to week 75
Population: SAS included all randomized participants exposed to at least one dose of randomized treatment.
Measure: Number; unit: Events
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 133 | 67
Events | 17 | 7

35. Secondary Outcome: Change in Pulse
Description: Change in pulse from baseline to week 68 is presented. Data is reported for on-treatment period: the on-treatment period was defined as the interval from first to last trial product administration plus 2 weeks of follow-up and excluding any period of temporary treatment interruption defined as >2 consecutive missed doses (corresponding to >2 weeks off-treatment).
Time Frame: Baseline (week 0), week 68
Population: SAS included all randomized participants exposed to at least one dose of randomized treatment. Overall Number of Participants Analyzed = number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Beats per minute (beats/min)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 119 | 58
Beats per minute (beats/min) | 0 (13) | -1 (13)

36. Secondary Outcome: Change in Amylase: Ratio to Baseline
Description: Change in amylase (U/L) from baseline to week 68 is presented as ratio to baseline. Data is reported for on-treatment period: the on-treatment period was defined as the interval from first to last trial product administration plus 2 weeks of follow-up and excluding any period of temporary treatment interruption defined as >2 consecutive missed doses (corresponding to >2 weeks off-treatment).
Time Frame: Baseline (week 0), week 68
Population: SAS included all randomized participants exposed to at least one dose of randomized treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of amylase
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 133 | 67
Ratio of amylase | 1.15 (17.4) | 1.04 (18.2)

37. Secondary Outcome: Change in Lipase: Ratio to Baseline
Description: Change in lipase (U/L) from baseline to week 68 is presented as ratio to baseline. Data is reported for on-treatment period: the on-treatment period was defined as the interval from first to last trial product administration plus 2 weeks of follow-up and excluding any period of temporary treatment interruption defined as >2 consecutive missed doses (corresponding to >2 weeks off-treatment).
Time Frame: Baseline (week 0), week 68
Population: SAS included all randomized participants exposed to at least one dose of randomized treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of lipase
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 133 | 67
Ratio of lipase | 1.39 (37.3) | 1.12 (37.0)

38. Secondary Outcome: Change in Calcitonin: Ratio to Baseline
Description: Change in calcitonin (nanograms per liter [ng/L]) from baseline to week 68 is presented as ratio to baseline. Data is reported for on-treatment period: the on-treatment period was defined as the interval from first to last trial product administration plus 2 weeks of follow-up and excluding any period of temporary treatment interruption defined as >2 consecutive missed doses (corresponding to >2 weeks off-treatment).
Time Frame: Baseline (week 0), week 68
Population: as for outcome 35
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of calcitonin
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 116 | 55
Ratio of calcitonin | 1.14 (47.0) | 1.09 (36.7)

ADVERSE EVENTS:
Time Frame: From baseline (week 0) to week 75
Description: All AEs reported here are TEAEs. TEAE is defined as an event that had onset date during the on-treatment period. The on-treatment period was defined as the interval from first to last trial product administration plus 7 weeks of follow-up and excluding any period of temporary treatment interruption defined as >7 consecutive missed doses (corresponding to >7 weeks off-treatment). SAS included all randomized participants exposed to at least one dose of randomized treatment.
Groups:
- Semaglutide 2.4 mg: Participants received once weekly s.c. injection of semaglutide for 68 weeks. Participants initially received 0.25 mg of semaglutide and the dose was then escalated once in 4 weeks for 16 weeks until the target dose of 2.4 mg was reached which was maintained for a period of 52 weeks: 0.25 mg (week 1 to week 4), 0.5 mg (week 5 to week 8), 1.0 mg (week 9 to week 12), 1.7 mg (week 13 to week 16) and 2.4 mg (week 17 to week 68). The treatment was an adjunct to a reduced-calorie diet and increased physical activity.
Arm/Group | Semaglutide 2.4 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/133 | 0/67
Serious Adverse Events (participants affected / at risk) | 15/133 | 6/67
Other Adverse Events (participants affected / at risk) | 90/133 | 40/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 2.4 mg (N=133) | Placebo (N=67)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 3 (3) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Post procedural constipation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 1 (1)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 2.4 mg (N=133) | Placebo (N=67)
Abdominal pain (Gastrointestinal disorders) | 20 (31) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 11 (19) | 8 (11)
Acne (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 4 (4)
COVID-19 (Infections and infestations) | 15 (16) | 10 (10)
Constipation (Gastrointestinal disorders) | 8 (8) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 8 (8) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 29 (54) | 13 (19)
Dizziness (Nervous system disorders) | 10 (13) | 2 (3)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 (3) | 4 (7)
Fatigue (General disorders) | 4 (4) | 5 (5)
Gastroenteritis (Infections and infestations) | 9 (9) | 2 (2)
Headache (Nervous system disorders) | 22 (52) | 11 (20)
Nasopharyngitis (Infections and infestations) | 16 (21) | 7 (12)
Nausea (Gastrointestinal disorders) | 56 (127) | 12 (29)
Pyrexia (General disorders) | 5 (5) | 5 (5)
Vomiting (Gastrointestinal disorders) | 48 (105) | 7 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-02-03): https://cdn.clinicaltrials.gov/large-docs/89/NCT04102189/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/89/NCT04102189/SAP_001.pdf